CLINICAL TRIAL: NCT06457256
Title: Hybrid Effectiveness-Implementation Trial of a School Clinician Training and Psychosocial ADHD/ODD Intervention Program Adapted for Schools Across Mexico (CLS-A-FUERTE)
Brief Title: Hybrid Effectiveness-Implementation Trial of a School Clinician Training and Psychosocial ADHD/ODD Intervention Program Adapted for Schools Across Mexico
Acronym: (CLS-A-FUERTE)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CLS-A-FUERTE
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: School Services as Usual (SAU) waitlist design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLS-A-FUERTE (Experimental): Receiving the CLS-A-FUERTE program immediately
  Interventions: Behavioral: CLS-A-FUERTE
- School Services as Usual (SA) (No Intervention): Receiving School Services as Usual while waiting to receive the CLS-A-FUERTE program in the subsequent schoolyear

INTERVENTIONS:
Behavioral: CLS-A-FUERTE — CLS-A-FUERTE Intervention Description: The CLS-A-FUERTE program is a school clinician training and psychosocial intervention program designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). Participating school clinicians are supported by a clinical research team of trainers who co-leads weekly training/consultation meetings and observes each intervention component (i.e., 6 weekly parent and student skills groups, as well as classroom management in the form of a Daily Report Card) in-vivo via videoconferencing.
  Arms: CLS-A-FUERTE

SUMMARY:
Neurodevelopmental disorders of Attention-Deficit/ Hyperactivity Disorder (ADHD) and Oppositional Defiant Disorder (ODD) are extremely common but underserved with Evidence- Based Treatments (EBT) worldwide. Thus, a school clinician training and ADHD/ODD intervention (i.e., the Collaborative Life Skills [CLS] program) was developed, implemented and evaluated for Mexico: a setting with high unmet need. Technology was integrated into the in-person program (CLS-FUERTE) to create a digitally enhanced version (CLS-R-FUERTE). Given findings demonstrating feasibility, acceptability, and efficacy of both program versions, a Type 2 Hybrid Effectiveness-Implementation Design will be applied to evaluate the program effectiveness, mechanisms of intervention change, and maintenance barriers/facilitators in a scaled-up cluster randomized controlled trial across two Mexican states -while simultaneously exploring an implementation strategy in which the program is adapted to enhance maintenance given each school's needs/resources (i.e., CLS-A-FUERTE). The implementation process is guided by the Exploration, Preparation, Implementation, and Sustainment (EPIS) model with evaluation following the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) Framework.

DETAILED DESCRIPTION:
Aim 1) Test the effectiveness and implementation of the CLS-A-FUERTE school clinician training and ADHD/ODD intervention program adapted for schools across Mexico. It is predicted:

H1) School clinicians will engage in training and implement chosen intervention components with fidelity H2) Teachers and/or families will engage in chosen intervention components and adhere to the strategies H3) Students receiving the CLS-A-FUERTE intervention will show greater improvements in ADHD/ODD symptoms and associated impairment compared to students receiving school services as usual

Aim 2) Evaluate mechanisms of sustained intervention change. It is predicted:

H4) Improvements in parenting behaviors will mediate sustained intervention effects H5) Improvements in teacher and/or school clinician competency will mediate intervention effects

Aim 3) Identify CLS-A-FUERTE maintenance barriers and facilitators. It is predicted that sustained intervention effects and continuation of program activities at follow-up will relate to:

H6) Program feasibility (i.e., cost estimates) and acceptability (i.e., participant satisfaction) H7) Characteristics of participating schools and school context factors

Aim 4) Expand research capacity to a novel university setting. It is predicted that emerging investigators will:

H8) Complete clinical research coursework and produce deliverables (i.e., presentations, papers, grants) H9) Show improved EBT skills, research capacity and culture ratings, and competency as program trainers

ELIGIBILITY:
Inclusion Criteria:

* must demonstrate at least six inattention symptoms and/or six hyperactive/impulsive symptoms endorsed by parent or teacher as occurring often or very often, AND at least one area of impairment rated as concerning by both parent and teacher, AND have a parent and teacher agreeing to participate (for student participants)
* Must be a parents, teacher, or school clinicians of participating students (for parent, teacher, and school clinician participants)
* Must be a university student in psychology or education at UAS or BUAP (for emerging investigator/university student participants)

Exclusion Criteria:

* inability to speak and read Spanish
* unstable medication regimen (for student participants)
* severe visual or hearing impairment (for student participants)
* severe language delay (for student participants)
* psychosis (for student participants)
* Placement in an all-day special education classroom (for student participants)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 872 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Child Symptom Inventory-4 (CSI-4) Parent Checklist ADHD Combined type Symptom Severity Score | Baseline and post treatment (8 weeks) and follow-up (3 months)
  Parents will assess ADHD symptoms using the CSI-4. The CSI-4: Parent Checklist contains 18 symptoms for ADHD, Combined type (ADHD:C; 18 items). Each symptom is rated on a 4-point scale (0= never to 3= very often). The average of ADHD:C scores range from zero to four, with higher scores indicating more severe symptoms.
Change in Child Symptom Inventory-4 (CSI-4) Teacher Checklist ADHD Combined type Symptom Severity Score | Baseline and post treatment (8 weeks) and follow-up (3 months)
  Teachers will assess ADHD symptoms using the CSI-4. The CSI-4: Teacher Checklist contains 18 symptoms for ADHD, Combined type (ADHD:C; 18 items). Each symptom is rated on a 4-point scale (0= never to 3= very often). The average of ADHD:C scores range from zero to four, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Change in Child Symptom Inventory-4 (CSI-4) Parent Checklist (Oppositional Defiant Disorder) ODD Symptom Severity Score | Baseline and post treatment (8 weeks) and follow-up (3 months)
  Parents will assess ODD symptoms using the CSI-4. The CSI-4: Parent Checklist contains 9 symptoms of ODD. Each symptom is rated on a 4-point scale (0= never to 3= very often). The average ODD scores range from zero to four, with higher scores indicating more severe symptoms.
Change in Child Symptom Inventory-4 (CSI-4) Teacher Checklist (Oppositional Defiant Disorder) ODD Symptom Severity Score | Baseline and post treatment (8 weeks) and follow-up (3 months)
  Teachers will assess ODD symptoms using the CSI-4. The CSI-4: Teacher Checklist contains 9 symptoms of ODD. Each symptom is rated on a 4-point scale (0= never to 3= very often). The average ODD scores range from zero to four, with higher scores indicating more severe symptoms.
Change Impairment Rating Scale (IRS) Parent Questionnaire Overall Severity Score | Baseline and post treatment (8 weeks) and follow-up (3 months)
  Parents will assess impairment using the IRS. The IRS Parent Questionnaire contains 8 items of functional impairment (i.e., academic and peer relations). Each item is rated on a 7-point scale (1= no problem; does not need treatment/services to 7= extreme impairment; definitely needs treatment/services). The average of all IRS scores range from one to seven, with higher scores indicating more severe impairment.
Change Impairment Rating Scale (IRS) Teacher Questionnaire Overall Severity Score | Baseline and post treatment (8 weeks) and follow-up (3 months)
  Teachers will assess impairment using the IRS. The IRS Teacher Questionnaire contains 8 items of functional impairment (i.e., academic and peer relations). Each item is rated on a 7-point scale (1= no problem; does not need treatment/services to 7= extreme impairment; definitely needs treatment/services). The average of all IRS scores range from one to seven, with higher scores indicating more severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Haack, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- UCSF, San Francisco, California, United States
- Mexico (2):
  - Benemérita Universidad Autónoma de Puebla, Puebla City, Puebla
  - Universidad Autonoma de Sinaloa, Culiacán, Sinaloa

IPD SHARING:
Plan to Share IPD: No